CLINICAL TRIAL: NCT02966470
Title: Hand Grip Strength as a Marker of Frailty in Surgical Patients
Status: Terminated | Type: Observational
Why Stopped: Due to accrual not met and PI no longer at the institution
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1609018398
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Frailty
Keywords: surgical outcomes
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General surgery patient: General surgery patient admitted to the Section of General Surgery, Trauma, and Surgical Critical Care who are over 60.
  Interventions: Device: Obtain grip strength from a standardized gripometer

INTERVENTIONS:
Device: Obtain grip strength from a standardized gripometer — Obtain grip strength from a standardized gripometer, 3 times on each hand

SUMMARY:
This study aims to assess if grip strength can be used as a single, objective surrogate of frailty assessment in the surgical population.

DETAILED DESCRIPTION:
Frailty is associated with worse outcomes. Current screening surveys are cumbersome, most containing multiple components. For frail patients particularly, it can be difficult to ascertain all the information requested. There is a need for a simple, one step, objective screening measure of frailty. There is some evidence in the medicine patients that grip strength may be related to frailty, but no such information is available for surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* General surgery patient admitted to the Section of General Surgery, Trauma, and Surgical Critical Care
* Age >60

Exclusion Criteria:

* Pregnancy
* Untreated or metastatic malignancy
* Prisoners

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General surgery patients admitted to the Section of General Surgery, Trauma, and Surgical Critical Care who are over the age of 60.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
linear regression of grip strength to frailty survey score | 10 minutes at the time of admission
  Their frailty survey and grip strength scores will also be recorded for analysis.
  We will analyze the data by linear regression of grip strength to frailty survey score.

CONTACTS AND LOCATIONS:
Overall Officials: Bishwajit Bhattacharya, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No